CLINICAL TRIAL: NCT03635216
Title: The Biomarker Analysis in Locally Advanced Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Jen Chen, Chair, Mackay Memorial Hospital
Other Study IDs: 18MMHIS060e
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Cervical cancer; Biomarker; Recurrence
MeSH Terms: conditions — Uterine Cervical Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — cervical cancer specimen for immunohistochemistry staining
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sonic hedgehog (Shh) signaling, including Gli1, is critical to treatment resistance. For optimizing cervical cancer treatment, the pathological prognostic factors determine whether to administer adjuvant therapy. However, the majority of clinical results was from squamous cell carcinoma, rendering conclusions for adenocarcinoma less convincing. We aimed to examine the role of Shh signaling in long-term clinical outcomes of cervical adenocarcinoma after receiving major surgery.

DETAILED DESCRIPTION:
Surgery, radiotherapy, and chemotherapy could achieve favorable locoregional control in cervical cancer. Although good local control results, distant failure plays a major role in patients with treatment failure.

We were interested in the potential biomarkers for recurrence after primary treatment for the following reasons. We wanted to identify patients at a high risk of recurrence. Such patients must be intensively monitored. We required baseline data, such as the actuarial relapse rate, for evaluation in an additional randomized study. Hence, we retrospectively analyzed the potential biomarkers for recurrence in cervical cancer. Statistical analysis of the data was done using the chi-square test. Disease free survival curves were constructed using the Kaplan-Meier method. Comparisons between curves were performed using the log-rank test. Multivariate analyses of factors associated with local and distant failure were made by logistic regression analysis.

From 1987 to 2002, 62 patients with cervical adenocarcinoma that received major surgery were enrolled for analysis of Shh signaling with a median follow-up period for 172.6 months (IQR 33.0-226.2 months). External beam radiotherapy with 50-60 Gy followed by brachytherapy with 30 Gy was delivered with or without concurrent weekly cisplatin 40 mg/m2. Clinical outcomes in terms of local recurrence, progression free survival (PFS) and overall survival (OS) will be analyzed. The expressions of Shh, Ptch-1, Smo and Gli1 were assessed by immunohistochemistry. Statistics will be performed using International Business Machines (IBM) Statistical Package for the Social Science (SPSS) v22.

ELIGIBILITY:
Inclusion Criteria:

* cervical cancer patients
* performance status Eastern Cooperative Oncology Group 0-1 (ECOG 0-1)

Exclusion Criteria:

* non-other cancer previously

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — cervical cancer only occurring in women
Study Population: Patients with cervical adenocarcinoma that received major surgery. External beam radiotherapy with 50-60 Gy followed by brachytherapy with 30 Gy was delivered with or without concurrent weekly cisplatin 40 mg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
Shh, Ptch-1, Smo and Gli1 | 1987-2002
  Sonic hedgehog (Shh) signaling, including Gli1, is critical to treatment resistance. to examine the role of Shh signaling in long-term clinical outcomes of cervical adenocarcinoma after receiving major surgery

SECONDARY OUTCOMES:
overall survival | 1987-2002
  The length of time from either the date of diagnosis or the start of treatment for cervical cancer
progression free survival | 1987-2002
  the length of time during and after the treatment of cervical cancer
local recurrence | 1987-2002
  cervical cancer that has recurred at or near the same place as the original tumor

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jen Chen, MD, Study Chair — Department of Radiation Oncology, MacKay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hong JH, Tsai CS, Chang JT, Wang CC, Lai CH, Lee SP, Tseng CJ, Chang TC, Tang SG. The prognostic significance of pre- and posttreatment SCC levels in patients with squamous cell carcinoma of the cervix treated by radiotherapy. Int J Radiat Oncol Biol Phys. 1998 Jul 1;41(4):823-30. doi: 10.1016/s0360-3016(98)00147-3. PMID 9652844
- [Background] Ogino I, Nakayama H, Kitamura T, Okamoto N, Inoue T. The curative role of radiotherapy in patients with isolated para-aortic node recurrence from cervical cancer and value of squamous cell carcinoma antigen for early detection. Int J Gynecol Cancer. 2005 Jul-Aug;15(4):630-8. doi: 10.1111/j.1525-1438.2005.00119.x. PMID 16014117
- [Background] Huang EY, Wang CJ, Chen HC, Fang FM, Huang YJ, Wang CY, Hsu HC. Multivariate analysis of para-aortic lymph node recurrence after definitive radiotherapy for stage IB-IVA squamous cell carcinoma of uterine cervix. Int J Radiat Oncol Biol Phys. 2008 Nov 1;72(3):834-42. doi: 10.1016/j.ijrobp.2008.01.035. Epub 2008 Apr 24. PMID 18439764